CLINICAL TRIAL: NCT04685239
Title: Risk of Dislocation After Total Hip Replacement: Dual Mobility Cup vs. Unipolar Cup. A Randomized Controlled Trial With Patients ≥65 Years Operated for Hip Osteoarthritis With Primary Total Hip Replacement (THR).
Brief Title: Dual Mobility Cup Versus Unipolar Cup
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20190040
Record Dates: First submitted 2020-12-15; First posted 2020-12-28 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Dislocation, Hip
Keywords: dislocation, hip; thr; dual mobility cup
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Intervention Model Description: controlled randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unipolar cup (Active Comparator): Patients randomized to receive a conventional unipolar acetabular cup
  Interventions: Device: unipolar cup
- dual mobility cup (Active Comparator): Patients randomized to receive a double mobility acetabular cup
  Interventions: Device: dual mobility cup

INTERVENTIONS:
Device: dual mobility cup — The use of a Sunfit dual mobility cup
  Arms: dual mobility cup
Device: unipolar cup — The use of a TMT cup
  Arms: Unipolar cup

SUMMARY:
The general purpose of this study is to examine whether the dual mobility cup (Novae® Serf) reduces the number of hip dislocations after total hip replacement, both early dislocation (≤1 year) and late dislocation (>1 year) after primary THR compared with a conventional cup design (Trabecular MetalTM Modular Acetabular System).

DETAILED DESCRIPTION:
Surgery with THR for arthritis and other hip disorders has long been one of the most successful orthopedic surgical treatments. The majority of the patients gain pain relief and experience improved hip function. In 2017, a total of 10,691 THRs were implanted in Denmark (annual report 2018).

Hip dislocation is a known complication after THR. It is a painful condition which may have far-reaching consequences for the patient, who may experience both physical and mental discomfort. Ultimately, multiple hip dislocations may result in reoperation.

In the literature, the incidence of hip dislocation is reported at 2-6 %, and a more recent review reports a risk of 0.5-10 %.

In Denmark, recurrent hip dislocation is the cause of 21 % of the reoperations per year according to The Danish Hip Arthroplasty Register. According to the British National Joint Registry (NJR) and the Australian register (AOANJRR), hip dislocation is the cause of 15.5 % and 21 %, respectively, of the reoperations.

The best method to avoid reoperation due to instability is to choose the correct implant for the individual patient and thereby spare the patient of having to endure a painful complication and yet another procedure. There are multiple risk factors for instability after THR, and increased use of dual mobility cups (DMC) is already documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip arthritis who are amenable to surgery with THR and age ≥ 65 years referred to the Department of Orthopedic Surgery at either Section Farsø, Frederikshavn Hospital or Aalborg University Hospital. Patients who are willing to participate in the trial and who give their written, informed consent after receiving oral and written information.

Exclusion Criteria:

* Patients who do not wish to participate.
* Sequelae of Calvé-Legg-Perthes' disease, caput necrosis, epiphysiolysis.
* Proximal femoral or acetabular fracture.
* Hip dysplasia with subluxation Crowe types III and IV.
* Earlier hip bone surgery (excluding arthroscopic surgery).
* Elective bilateral surgery.
* If the patient's bone morphology is unsuitable for a cemented Exeter® femoral stem.
* Patients with no e-mail.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Early dislocation, Difference in dislocation within 1 year. | 1 year after surgery
  The primary outcome is the difference in cumulative incidence proportion of dislocation between the 2 randomized groups within the first year after total hip replacement. The information will be collected from both the patient through questionnaires and from the Danish Hip Arthroplasty Register and the Danish National Patient Register.

SECONDARY OUTCOMES:
Difference in dislocation within 5 years | 5 years after surgery
  The difference in cumulative incidence proportion of dislocation between the 2 randomized groups within 5 years after total hip replacement. The information will be collected from both the patient through questionnaires and from the Danish Hip Arthroplasty Register and the Danish National Patient Register.
Dislocation 10 year | 10 years after surgery
  The difference in cumulative incidence proportion of dislocation between the 2 randomized groups within 10 years after total hip replacement. The information will be collected from both the patient through questionnaires and from the Danish Hip Arthroplasty Register and the Danish National Patient Register.
Prosthesis survival. | 1, 5 and 10 year
  Evaluated by the cumulative incidence of THR's reoperated within 1, 5 and 10 years after total hip replacement. The information will be collected from both the patient through questionnaires and from the Danish Hip Arthroplasty Register and the Danish National Patient Register.
Patient reported outcome measure: European quality of life 5 dimensions (EQ-5D 5L) | 1, 5 and 10 years
  Patients will be scored with EQ-5D 5L preoperatively and at 1,5 and 10 years. It consists of 5 dimensions ranging from 1-5, with 1 being the best in each dimension. It also consist of a visual analog scale ranging from 0-100, 100 being the best imaginable health, The EQ VAS describes the respondents current overall health. Data will be showed as changes in health over time showing responses at baseline and at follow up or as frequencies and proportions reported by dimension and level.
Patient reported outcome measure: Oxford Hip Score (OHS) | 1, 5 and 10 years
  Patients will be scored with OHS at baseline and at 1, 5 and 10 years. OHS is a patient-recorded outcome measure designed to assess the outcome of hip replacements. Its a score between 0-48 with 48 being the best.
Patient reported outcome measures: The Copenhagen Hip and Groin Outcome Score (HAGOS) | 1, 5 and 10 years
  HAGOS pain subscale will be used to report pain pre and postoperatively. The score in the pain subscale ranges from 0 (extreme hip/groin problems) -100 (no hip/groin problems).

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, Northen Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No